CLINICAL TRIAL: NCT01271829
Title: Incorporating Avocados in Meals: Effect on Glycemic Index, Insulin Response, Satiety and Satiety-related Gastrointestinal Peptides in Humans
Brief Title: Incorporating Avocados in Meals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: Hass Avocado Board (Other)
Responsible Party: Principal Investigator, Joan Sabate,DrPH, MD, Chair, Department of Nutrition, Loma Linda University
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 5100220
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Satiety; Glycemic Index; Insulin; Gastrointestinal Peptides and Hormones
Keywords: Avocados; Satiety; Feeding study
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): While on the control arm subjects will be given a meal with no avocado.
- Avocado supplement (Active Comparator): While on the avocado supplement arm subjects will be given a meal in which a given amount of calories will be replaced by calories contributed by avocados.
  Interventions: Dietary Supplement: Avocado supplement
- Avocado included (Active Comparator): While on the avocado included arm subjects will be given a meal in which the calories of avocado will be added to the calories of the control meal.
  Interventions: Dietary Supplement: Avocado included

INTERVENTIONS:
Dietary Supplement: Avocado supplement — Calories from avocados replace calories of the control lunch
  Arms: Avocado supplement
Dietary Supplement: Avocado included — Calories from avocados will be added to calories from the control lunch
  Arms: Avocado included

SUMMARY:
The purpose of this study is to examine the effect of incorporating avocados in meals on post-ingestion glycemic index, insulin response, sensations of satiety and on appetite-related gastrointestinal peptide and hormone release. Also the effect of consuming avocado containing meals on the caloric intake of participants in subsequent eating episodes will be explored.

Each subject will participate in one intervention for one day, wait one or two weeks, come for another intervention, wait one or two weeks and come for a final intervention- three in total. Participants will be randomly assigned to one of six treatment sequences. Postprandial response to the control and two avocado-containing test meals will be assessed and compared using a 3 x 3 single blind cross-over design. The Subjects will be between 25 and 60 years old, female or male, with a BMI of 23 to 32, stable weight, no sports involvement, non-smoking and not dependent on caffeine. Thirty subjects will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* 23-60 years old
* BMI 23-32
* Stable weight for 6 months
* Live or work near Loma Linda University

Exclusion Criteria:

* Smoker
* Heavy involvement in sports
* Dependent on caffeine

Ages: 23 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Satiety | 12 hours
  The effect that consumption of avocados has on feelings of fullness and the quantity of food consumed in a subsequent eating episode

SECONDARY OUTCOMES:
post-ingestion glycemic index | 3 hours
  Blood will be drawn at 30 minutes, 60 minutes, 120 minutes and 180 minutes after consumption of a meal with or without avocados. The glycemic index will be analyzed.
insulin response | 3 hours
  Blood will be drawn at 30 minutes, 60 minutes, 120 minutes and 180 minutes after consumption of a meal with or without avocados. Insulin response will be analyzed.
appetite-related gastrointestinal peptide and hormone release | 3 hours
  Blood will be drawn at 30 minutes, 60 minutes, 120 minutes and 180 minutes after consumption of a meal with or without avocados. Gastrointestinal peptide and hormones will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Sabaté, MD, DrPH, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Department of Nutrition, Loma Linda, California, United States

REFERENCES:
- [Result] Wien M, Haddad E, Oda K, Sabate J. A randomized 3x3 crossover study to evaluate the effect of Hass avocado intake on post-ingestive satiety, glucose and insulin levels, and subsequent energy intake in overweight adults. Nutr J. 2013 Nov 27;12:155. doi: 10.1186/1475-2891-12-155. PMID 24279738
- See also: Publication of study results — http://www.nutritionj.com/content/12/1/155